CLINICAL TRIAL: NCT03403036
Title: A Study to Evaluate the Safety and Efficacy of Brodalumab in Subjects With Moderate to Severe Plaque Psoriasis Who Have Failed IL-17A Therapies
Brief Title: Brodalumab in Subjects With Moderate to Severe Plaque Psoriasis Who Have Failed IL-17A Therapies
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Mark Lebwohl, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 17-1581
Record Dates: First submitted 2018-01-11; First posted 2018-01-18 (Actual); Results first posted 2019-07-09 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-02

CONDITIONS: Psoriasis
Keywords: Psoriasis; brodalumab
MeSH Terms: conditions — Psoriasis | interventions — brodalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Brodalumab (Experimental): Brodalumab (210 mg) via subcutaneous injection using prefilled syringes
  Interventions: Drug: Brodalumab

INTERVENTIONS:
Drug: Brodalumab — Weeks 0, 1, 2, and every 2 weeks thereafter through and including Week 16.
  Other Names: Siliq

SUMMARY:
This study will evaluate the safety and efficacy of brodalumab in the treatment of moderate-to-severe psoriasis in patients who have previously failed treatment with interleukin (IL)-17A therapies. Forty patients will be enrolled in this 16-week open-label study. Patients will receive 210 mg of brodalumab subcutaneous injection at weeks 0, 1, and 2, followed by 210 mg every 2 weeks. The primary efficacy endpoint will be the proportion of patients achieving a score of "0-clear" or "1-almost clear" in the sPGA score after 16 weeks of treatment. After completion of the 16-week trial, patients may desire to continue treatment with brodalumab.

DETAILED DESCRIPTION:
This study will evaluate the safety and efficacy of brodalumab in the treatment of moderate-to-severe psoriasis in patients who have previously failed treatment with interleukin (IL)-17A therapies. Failure of IL-17A therapy will be defined as previous treatment with either secukinumab or ixekizumab for at least 3 months without achieving PASI-75 response or a 50% loss of original improvement. Forty patients will be enrolled in this 16-week open-label study. Patients will be enrolled at three to four different sites in the US. After enrollment, study visits will occur at monthly intervals, with patients receiving 210 mg of brodalumab subcutaneous injection at weeks 0, 1, and 2, followed by 210 mg every 2 weeks. At each visit, patients will be evaluated for change in sPGA (Physician's Global Assessment), PASI score, and any signs or symptoms of adverse events. Laboratory screening will include tests for tuberculosis and neutropenia. After completion of the 16-week trial, patients may desire to continue treatment with brodalumab. Efforts will be made to provide drug to these study patients, including those who do not have insurance.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject at least 18 years of age
* Subject is able to provide written informed consent and comply with the requirements of this study protocol.
* Have both a sPGA score of ≥3 and BSA ≥ 5% prior to randomization.
* Subjects who are women of childbearing potential must have a negative urine pregnancy test at screening and must be practicing an adequate, medically acceptable method of birth control for at least 30 days before Day 0 and at least 6 months after the last study drug administration. Acceptable methods of birth control include intrauterine device (IUD); oral, transdermal, implanted or injected hormonal contraceptives (must have been initiated at least 1 month before entering the study); tubal ligation; abstinence and barrier methods with spermicide. Otherwise, if not of childbearing potential, subjects must: have a sterile or vasectomized partner; have had a hysterectomy, a bilateral oophorectomy or be clinically diagnosed infertile; or be in a menopausal state for at least a year.
* Tuberculin purified protein derivative (PPD) or QuantiFERON TB-Gold test (QFT) negative at the time of screening, or if patient has a history of positive PPD or QuantiFERON, he/she has initiated or completed the appropriate prophylaxis.
* Subject is judged to be in good general health as determined by the principal investigator based upon the results of medical history and laboratory profile.
* Subject has previously failed treatment with an IL-17A agent, secukinumab or ixekizumab, (where available, defined as previous treatment with either drug for at least 3 months without achieving PASI-75 response or a 50% loss of original improvement).
* Last administration of secukinumab or ixekizumab ≥ 28 days prior to Baseline.

Exclusion Criteria:

* Have predominantly pustular, erythrodermic, and/or guttate forms of psoriasis.
* History of an ongoing, chronic or recurrent infectious disease, or evidence of tuberculosis infection as defined by a positive tuberculin purified protein derivative (PPD) or QuantiFERON TB-Gold test (QFT) at Screening. Subjects with a positive or indeterminate PPD or QFT test may participate in the study if a full tuberculosis work up (according to local practice/guidelines) is completed within 12 weeks prior to randomization and establishes conclusively that the subject has no evidence of active tuberculosis. If presence of latent tuberculosis is established, then treatment must have been initiated at least for 4 weeks prior to randomization and the course of prophylaxis is planned to be completed.
* Subjects with a history of HIV, or history of positive HCV or HBV
* Use of any of the following therapies within 4 weeks prior to Baseline (Visit 2): systemic non-biologic psoriasis therapies (including, but not limited to): psoralens and ultraviolet A (PUVA) therapy, cyclosporine, methotrexate, azathioprine, corticosteroids, apremilast, tofacitinib, oral retinoids, mycophenolate mofetil, sirolimus; 1, 25 dihydroxyvitamin D analogs; or phototherapy (including UVB or self-treatment with tanning beds or therapeutic sunbathing) or topical psoriasis therapy with psoralens.
* Use of topical corticosteroid preparations, topical calcineurin inhibitors, or other topical preparations with immunomodulatory properties within 2 weeks prior to Baseline (Visit 2).
* Use of any investigational drug or any systemic drug for psoriasis within four weeks prior to Baseline (Visit 2).
* Serious concomitant illness that could require the use of systemic corticosteroids or otherwise interfere with the patient's participation in the trial.
* Clinically important deviation as judged by the investigator (such WBC< 3) from normal limits in physical examination, vital sign measurements, clinical laboratory tests results, not associated with a chronic, well-controlled medical condition.
* Any active live-vaccines 3 months prior to baseline and throughout the study.
* Have a current or history of lymphoproliferative disease within 5 years prior to Baseline (Visit 2); or have current or history of any malignant disease within 5 years prior to Baseline (Visit 2).
* History of suicide attempt, or are clinically judged by investigator to be at risk of suicide.
* History of Crohn's disease.
* Had a serious infection, been hospitalized, or received IV antibiotics for an infection, within 12 weeks prior to Baseline (Visit 2).
* Known immunodeficiency, or history of infection typical of an immunocompromised host.
* At screening, have a neutrophil count <1500 cells/uL.
* At screening, have a lymphocyte count <800 cells/uL.
* At screening, have a platelet count <100,000 cells/uL.
* At screening, have a total white blood count (WBC) < 3000 cells/uL.
* At screening, have a hemoglobin <8.5 g/dL.
* Have donated >450 mL of blood within 4 weeks prior to screening (Visit 1), or intend to donate blood during the course of the study.
* Women who are lactating or breastfeeding.
* Any other condition that precludes the patient from following and completing the protocol, in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2017-10-31 (Actual); Primary Completion 2018-08-18 (Actual); Study Completion 2018-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Lebwohl, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Baylor College of Medicine, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 41 patients screened with 39 meeting all eligibility requirements. Patients with moderate-to-severe psoriasis were recruited from 3 sites.
Groups:
- Brodalumab: Brodalumab (210 mg) via subcutaneous injection using prefilled syringes given at Weeks 0, 1, 2, and every 2 weeks thereafter through and including Week 16.
Period: Overall Study
Arm/Group | Brodalumab
Started | 39
Completed | 34
Not Completed | 5
Not completed — Lack of Efficacy | 5

BASELINE CHARACTERISTICS:
Arm/Group | Brodalumab
Number analyzed (Participants) | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.74 (2.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 25
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Baseline PASI [Mean (Standard Deviation); unit: units on a scale] — Psoriasis Area and Severity Index (PASI) - combines the assessment of the severity of lesions and the area affected into a single total score in the range 0 (no disease) to 72 (maximal disease). Higher score indicates more severe psoriasis.
  units on a scale | 20.36 (2.24)
Baseline sPGA [Mean (Standard Deviation); unit: units on a scale] — static Physician's Global Assessment (sPGA) is a 6-point numerical scale ranging from 0 (clear) to 5 (very severe) to assess psoriasis severity at a given time point .
  units on a scale | 3.41 (0.08)
Number of participants who failed Secukinumab [Count of Participants; unit: Participants] | 16
Number of participants who failed Ixekizumab [Count of Participants; unit: Participants] | 19
Number of participants who failed both Secukinumab and Ixekizumab [Count of Participants; unit: Participants] | 4
Number of previously failed biologics [Mean (Standard Deviation); unit: biologic medications] — The average number of total failed biologic agents per patient
  biologic medications | 2.23 (0.29)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Physician's Global Assessment (sPGA) Score 0 or 1
Description: Number of patients achieving a score of "0-clear" or "1-almost clear" in the sPGA score after 16 weeks of treatment to measure efficacy.
  Static Physician Global Assessment (sPGA) - 3 categories induration, erythema, and scaling, scored 0-4, these 3 categories averaged giving total score from 0-4, with higher score indicating more symptoms.
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Brodalumab
Number analyzed (Participants) | 34
Participants | 24

2. Secondary Outcome: Number of Participants With Psoriasis Area and Severity Index (PASI) Score Improvement
Description: PASI combines the assessment of the severity of lesions and the area affected into a single score in the range 0 (no disease) to 72 (maximal disease). Number of participants with 75%, 90%, and 100% reduction in the PASI score, respectively, PASI-75, PASI-90, and PASI-100 who completed the trial at week 16.
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Brodalumab
Number analyzed (Participants) | 34
Participants
  PASI-75 | 26
  PASI-90 | 17
  PASI-100 | 11

3. Secondary Outcome: Number of Adverse Events
Description: Number of adverse events as a measure of safety
Time Frame: 16 weeks
Measure: Number; unit: events
Arm/Group | Brodalumab
Number analyzed (Participants) | 39
events | 6

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Brodalumab
All-Cause Mortality (participants affected / at risk) | 0/39
Serious Adverse Events (participants affected / at risk) | 0/39
Other Adverse Events (participants affected / at risk) | 6/39
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brodalumab (N=39)
Corneal Ulcer (Eye disorders) | 1 (1)
Tooth Abscess (Infections and infestations) | 1 (1)
Allergic Sinusitis (Immune system disorders) | 1 (1)
Folliculitis (Skin and subcutaneous tissue disorders) | 1 (1)
Pre-Diabetes (Endocrine disorders) | 1 (1)
Sciatica (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-12): https://cdn.clinicaltrials.gov/large-docs/36/NCT03403036/Prot_SAP_000.pdf